CLINICAL TRIAL: NCT04738539
Title: Efficacy of Contrast Enhanced Voiding Urosonography for Urodynamic Studies
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Nora Kern, MD, Associate Professor, Department of Urology, University of Virginia
Other Study IDs: HSR200346
Record Dates: First submitted 2021-02-01; First posted 2021-02-04 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Myelomeningocele; Neurogenic Bladder; Tethered Cord Syndrome; Bladder, Neurogenic; Urologic Diseases; Neurologic Dysfunction
Keywords: Contrast Enhanced Voiding Urosonography; Urodynamics; Neurogenic Bladder; Detrusor Sphincter Dyssynergia
MeSH Terms: conditions — Meningomyelocele; Urinary Bladder, Neurogenic; Neural Tube Defects; Urologic Diseases; Neurologic Manifestations | interventions — Urodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with or being evaluated for neurogenic bladder: Pediatric patients presenting to UVA Pediatric Urology for follow up or repeat urodynamics testing.
  Interventions: Drug: Contrast Enhanced Voiding Urosonography with Urodynamic Testing; Diagnostic Test: Urodynamic Testing

INTERVENTIONS:
Drug: Contrast Enhanced Voiding Urosonography with Urodynamic Testing — We will be using contrast enhanced voiding urosonography to image urodynamic testing on patients with neurogenic bladder.
  Other Names: CeVUS; Contrast Enhanced Voiding Urosonography
Diagnostic Test: Urodynamic Testing — We will be using contrast enhanced voiding urosonography to image urodynamic testing on patients with neurogenic bladder.
  Other Names: Urodynamics

SUMMARY:
The investigators will assess the feasibility of replacing fluoroscopy/iodinated contrast with ultrasound/sulfur hexafluoride lipid-type A microspheres during routine urodynamic studies.

DETAILED DESCRIPTION:
Urodynamic studies routinely involve instillation of iohexol (OmnipaqueTM), a low osmolality contrast agent, into the bladder followed by fluoroscopic imaging to assess for reflux or variant anatomy of the genitourinary system. Recently, sulfur hexafluoride lipid-type A microspheres (LumasonTM), an ultrasound contrast agent, has been approved in the United States for intravesicular administration in the pediatric population. Contrast enhanced voiding urosonography (CEvUS) is being increasingly utilized in the place of voiding cystourethrograms, with the major advantages being decreased (zero) radiation for the patient, as well as decreased cost. Given the similarity in procedure between urodynamic studies (UDS) and voiding cystourethrograms, we hypothesize that a urodynamic study may be performed with contrast enhanced ultrasound instead of fluoroscopy. We plan to continue enrollment from our feasibility study and perform an efficacy study by recruiting a group of 105 patients under the age of 18, who are willing to undergo their normally schedule UDS using CEvUS to image the study in place of fluoroscopy. The UDS typically consists of two cycles of bladder filling and voiding; we intend replace the use of fluoroscopy and iohexel with ultrasound and sulfur hexafluoride lipid-type A microspheres. This will decrease the time commitment and eliminate radiation exposure for the patient. Data to be analyzed will include images from the study and patient/caregiver preference. Results from the ceVUS images will be compared to images obtained during previous tests imaged with fluoroscopy from the same patients currently enrolled in this study. Bladder shape and morphology, bladder neck configuration and performance, structure of the urethra, presence and degree of vesicoureteral reflux, and active voiding images will all be compared to fluoroscopy images from previous studies. The purpose of the study is to demonstrate that ceVUS is effective as an imaging technique for urodynamic studies, with an ultimate goal of using ceVUS instead of fluoroscopy in all urodynamic and voiding studies in order to decrease pediatric radiation exposure. The hypothesis is that ceVUS will be as effective for imaging urodynamics studies as fluoroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17
* Must have had prior urodynamic study at UVA

Exclusion Criteria:

* Pregnant women (self-reported)
* Fetuses
* Neonates
* Prisoners
* Subjects with preexisting cardiac conditions (such as CHF and ventricular arrhythmias)
* Subjects with a known hypersensitivity to Lumason

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients presenting to UVA Pediatric Urology for follow up or repeat urodynamics study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-03-02 (Estimated); Study Completion 2022-03-02 (Estimated)

PRIMARY OUTCOMES:
Bladder shape and morphology | Procedure (At time of urodynamic investigation)
  Comparison of previous fluroscopy images and ceVUS images
Bladder neck configuration | Procedure (At time of urodynamic investigation)
  Comparison of previous fluroscopy images and ceVUS images
Structure of urethra | Procedure (At time of urodynamic investigation)
  Comparison of previous fluroscopy images and ceVUS images
Presence and degree of VUR | Procedure (At time of urodynamic investigation)
  Comparison of previous fluroscopy images and ceVUS images
Images of active voiding | Procedure (At time of urodynamic investigation)
  Comparison of previous fluroscopy images and ceVUS images

SECONDARY OUTCOMES:
Patient/caregiver preference | Immediately following urodynamic investigation or up to 7 days after by phone
  Comparison survey

CONTACTS AND LOCATIONS:
Overall Officials: Nora G Kern, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Drzewiecki BA, Bauer SB. Urodynamic testing in children: indications, technique, interpretation and significance. J Urol. 2011 Oct;186(4):1190-7. doi: 10.1016/j.juro.2011.02.2692. Epub 2011 Aug 16. PMID 21849190
- [Background] Fernbach SK, Feinstein KA, Schmidt MB. Pediatric voiding cystourethrography: a pictorial guide. Radiographics. 2000 Jan-Feb;20(1):155-68; discussion 168-71. doi: 10.1148/radiographics.20.1.g00ja12155. PMID 10682779
- [Background] Mane N, Sharma A, Patil A, Gadekar C, Andankar M, Pathak H. Comparison of contrast-enhanced voiding urosonography with voiding cystourethrography in pediatric vesicoureteral reflux. Turk J Urol. 2018 May;44(3):261-267. doi: 10.5152/tud.2018.76702. Epub 2018 Mar 6. PMID 29733800
- See also: Feasibility of Using Contrast Enhanced Voiding Urosonography (CeVUS) During Urodynamic Studies (NCT04170413) — https://www.clinicaltrials.gov/ct2/show/NCT04170413?term=lumason&cond=Neurogenic+Bladder&cntry=US&state=US%3AVA&city=Charlottesville&draw=2&rank=1